CLINICAL TRIAL: NCT06141330
Title: Vitamin D Supplementation in Combination With Azithromycin and Topical Retinoid for Acne: A Randomized Controlled Trial
Brief Title: Vitamin D Supplementation in Acne
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aqsa Naheed, Professor, MBBS, FCPS, HITEC-Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vit-D
Record Dates: First submitted 2023-10-23; First posted 2023-11-21 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Acne Vulgaris
Keywords: AcneVulgaris; Vitamin D
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D (Experimental)
  Interventions: Dietary Supplement: D Max Drops; Drug: Azithromycin 250 milligram Oral Capsule; Drug: Adapalene
- Placebo (Active Comparator)
  Interventions: Drug: Azithromycin 250 milligram Oral Capsule; Drug: Adapalene

INTERVENTIONS:
Dietary Supplement: D Max Drops — Vitamin D
  Arms: Vitamin D
Drug: Azithromycin 250 milligram Oral Capsule — Anti Biotic
Drug: Adapalene — Retinoid

SUMMARY:
The goal of this clinical trial is to compare in acne vulgaris patients. The main question it aims to answer is:

• To assess the therapeutic benefit of vitamin D supplement in acne vulgaris treatment, following a 2-month treatment regimen that includes vitamin D supplementation compared to conventional (systemic azithromycin and topical retinoid) treatment alone.

Participants will receive vitamin D supplements in addition to capsule Azithromycin and topical retinoid.

Researchers will compare groups to determine efficacy of Vitamin D supplements in the treatment of Acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 13 and 40 years with diagnoses of Acne vulgaris are included.

Exclusion Criteria:

* Individuals currently undergoing treatment for polycystic ovary syndrome (PCOs)
* Those with obesity
* Individuals employing vitamin supplementation
* Those under the influence of topical or systemic steroids and acne treatment in the last 2 months.

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-02-24 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Efficacious | 2 months
  Improvement in Global Acne Grading System Score from baseline to after 2 months of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hitec-Ims, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
not sharing